CLINICAL TRIAL: NCT05082636
Title: The Role of Programmed Death Ligand -1 (Pdl-1) in Lung Cancer
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Norhan Salah Abd-Elmawgoud, Teaching and Research Assistant, Assiut University
Other Study IDs: PDL-1 Lung Cancer
Record Dates: First submitted 2021-09-24; First posted 2021-10-19 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: 54 patients with early stage lung (stage I, II) cancer (Group 1) were selected from the Chest Department of Assiut University Hospital,
  Interventions: Other: Observational Study ( Tissue Biopsy )
- control: besides 36 healthy controls; who were clinically suspicious with chest masses and proven histopathologically to be negative cancer (Group 2).
  Interventions: Other: Observational Study ( Tissue Biopsy )

INTERVENTIONS:
Other: Observational Study ( Tissue Biopsy ) — control study includes a total of 90 subjects. Of them 54 patients with early stage lung (stage I, II) cancer (Group 1) were selected from the Chest Department of Assiut University Hospital, besides 36 healthy controls; who were clinically suspicious with chest masses and proven histopathologically to be negative cancer (Group 2).obtained by fiberoptic bronchoscopy

SUMMARY:
This study was designed to investigate the correlation of lung cancer tissue expression of both PDL-1-mRNA ,vitamin D receptor (VDR) and level of vit.D in sera of lung cancer patients.These three biochemical markers may interact and play a role in lung cancer progression.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death worldwide. In 2018, it represented 11.6% of total cancer cases and 18.4% of total cancer deaths, making it the most frequent cancer and cause of cancer death in men and women combined .In Egypt, Lung cancer represents the most lethal malignancy and the fourth most common cancer in men.It is relatively more common in men. This gender difference in incidence is mainly due to differences in tobacco smoking rates, as smoking represents the major risk factor of this disease.

Programmed cell death 1 (PD-1) (Entrez Gene: 29126) and its ligand, programmed cell death ligand-1 (PDL-1) are new members of the CD28/B7 stimulatory superfamily. They mediate a negative signal, which inhibits functioning and proliferation of T and B cells, and reduce interleukin-2(IL-2), IL-10, and interferon-γ secretions.This inhibitory pathway is closely related to tumor progression, it provides an immune escape for tumor cells through cytotoxic T-cell inactivation. It plays an important role in the microenvironment of the tumor progress.Expression of this gene in tumor cells is prognostic in many types of human malignancies.Interaction of this ligand with its receptor inhibits T-cell activation and cytokine production. During infection or inflammation of normal tissue, this interaction is important for preventing autoimmunity by maintaining homeostasis of the immune response with local immune tolerance to tumors.

The biologically active form of Vit D, namely calcitriol or 1,25-dihydroxy Vitamin D (1,25(OH)2D ), is generated when 25(OH)D is hydroxylated in the kidneys by the cytochrome 1-α- hydroxylase enzyme (CYP27B1) (RXR) Yet, Vit. D has controversial effects; it has been shown to induce apoptosis of cancer cells and likely to play a promising role in cancer therapy.Numerous studies have proposed a strong relationship between low serum Vit. D levels and increased risk of cancer, especially by the strongest evidence in breast and colorectal cancer.

The biological actions as anti-cancer effects of calcitriol are mostly exerted through genomic actions mediated by the VDR and its existence in the numerous tumor tissues is suggestive of its role in tumor genesis.The VDR is a member of the nuclear receptor/steroid hormone receptor superfamily. These receptors function as ligand-activated, transcriptional regulatory proteins.VDR/RXR complex translocates into the nucleus and induces the transcription of phosphoinositide phospholipase C-γ1 (PLC-γ1) through interaction with Vit.D responsive element (VDRE) on specific genes.

There is an up-regulation of VDR upon exposure to Vit.D. The anti-proliferative and pro differentiating effects of Vit.D are mostly mediated through the nuclear VDR.In many types of cancers, decreased VDR expression has been found in advanced neoplasms.It was demonstrated a differential expression of VDR (nuclear/cytoplasm) in progression of normal to invasive squamous cell carcinoma.

In this study, we aimed to detect tissue PDL-1, VDR expression levels and serum Vit.D levels as biomarkers for the early detection of LC, investigating the correlations between these biochemical indices and the clinicopathological features, and different risk factors in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed histopathologically proven stage I and II lung cancer.

Exclusion Criteria:

* : patients who have pulmonary secondaries or metastasis (usually multiple and widespread tumors), and who received treatment for lung cancer or those suffering from other malignancies elsewhere were excluded from the current study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The mean age ±S.E for controls was 55.47 ± 1.5 year, while that of lung cancer cases was 56.31 ± 0.83 years.
  All patients were subjected to a full history taking, physical examination, routine laboratory investigations as blood picture, liver function, chest x- rays, chest ultrasonography. For patients who had been suspected clinically to have lung cancer, by examining the lung tissue obtained by fiberoptic bronchoscopic, the final diagnosis was confirmed histopathologically.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
measuring expression of PDL-1,VDR in cancer patients and healthy control. | through study completion, an average of 1 year.
  we measured PDL-1 and VDR expressions by real time q-PCR, in lung cancer tissues from patients with stage I and II LC and healthy controls who were clinically suspicious with chest masses and proven histopathologically to be negative cancer .

SECONDARY OUTCOMES:
measuring serum Vit D level by EIA method | through study completion, an average of 1 year.
  The level of serum Vitamin D (Vit.D) were assessed by EIA method.in lung cancer tissues from patients with stage I and II LC and healthy controls who were clinically suspicious with chest masses and proven histopathologically to be negative cancer .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Ceeraz S, Nowak EC, Noelle RJ. B7 family checkpoint regulators in immune regulation and disease. Trends Immunol. 2013 Nov;34(11):556-63. doi: 10.1016/j.it.2013.07.003. Epub 2013 Aug 13. PMID 23954143
- [Background] Zhang Y, Jiang X, Li X, Gaman MA, Kord-Varkaneh H, Rahmani J, Salehi-Sahlabadi A, Day AS, Xu Y. Serum Vitamin D Levels and Risk of Liver Cancer: A Systematic Review and Dose-Response Meta-Analysis of Cohort Studies. Nutr Cancer. 2021;73(8):1-9. doi: 10.1080/01635581.2020.1797127. Epub 2020 Jul 24. PMID 32705896
- [Background] Kim SH, Chen G, King AN, Jeon CK, Christensen PJ, Zhao L, Simpson RU, Thomas DG, Giordano TJ, Brenner DE, Hollis B, Beer DG, Ramnath N. Characterization of vitamin D receptor (VDR) in lung adenocarcinoma. Lung Cancer. 2012 Aug;77(2):265-71. doi: 10.1016/j.lungcan.2012.04.010. Epub 2012 May 6. PMID 22564539